CLINICAL TRIAL: NCT06546904
Title: Evaluation of the Effectiveness of Artificial Intelligence Empowered Ultrasound in Regional Anesthesia Training
Brief Title: Artificial Intelligence Empowered Anesthesia Ultrasound Guided Regional Anesthesia Training
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, aijun xu, Clinical Professor, Tongji Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: AISR
Record Dates: First submitted 2024-08-03; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Ultrasound-guided Regional Anesthesia
Keywords: artificial intelligence; ultrasound-guided regional anesthesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI group (Experimental): Group AI used artificial intelligence to empower anesthesia ultrasound assisted simulated PNB operations in 5 areas
  Interventions: Device: Artificial intelligence empowers anesthesia with ultrasound assistance
- Control group (No Intervention): Control group did not use AI assisted simulated PNB operations in 5 areas

INTERVENTIONS:
Device: Artificial intelligence empowers anesthesia with ultrasound assistance — Artificial intelligence empowers anesthesia with ultrasound assistance
  Arms: AI group

SUMMARY:
Evaluate the effectiveness of AI powered anesthesia ultrasound in ultrasound-guided regional anesthesia (UGRA) training.

DETAILED DESCRIPTION:
The AI powered anesthesia ultrasound system integrates ScanNav and NeedleTrainer modules, providing real-time training for medical staff to simulate punctures. Combined with ScanNav's real-time anatomical structure recognition function, it is expected to significantly enhance the training effectiveness of ultrasound-guided regional anesthesia technology.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participants;
* Sign the informed consent form.

Exclusion Criteria:

* allergic to ultrasound coupling agents

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Success rate of ultrasound-guided puncture | 1day
  Success rate of ultrasound-guided puncture at the first attempt

SECONDARY OUTCOMES:
Location time | 1day
  the time from the placement of the US transducer on the skin to the time of piercing of the skin.

CONTACTS AND LOCATIONS:
Overall Officials: mujun Chang, Dr., Study Chair — Tongji Hospital
Locations (1):
- Tongji hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No